CLINICAL TRIAL: NCT04814550
Title: Angiography-Derived Fractional Flow Reserve for Functional Evaluation of Coronary Artery Disease
Brief Title: Diagnostic Accuracy of CFD-Based Fractional Flow Reserve Derived From Coronary Angiography
Acronym: ACCURATE
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-153
Record Dates: First submitted 2020-12-06; First posted 2021-03-24 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FFR — FFR measured by pressure wire, AccuFFRangio computed by coronary angiographic images
  Other Names: AccuFFRangio

SUMMARY:
This is a prospective, multicenter, self-control clinical trial designed to assess the efficacy of AccuFFRangio, a novel method for evaluating the functional significance of coronary stenosis from coronary angiography, with FFR as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Stable or unstable angina, or myocardial infarction after the acute phase, indication for FFR in at least one vessel;
* Able to provide informed consent.

Exclusion Criteria:

* Subjects judged unsuitable for diagnostic intervention or FFR;
* Myocardial infarction within 6 days;
* LVEF ≤50%;
* eGFR <60ml/min（1.73m²）
* Severe coagulation dysfunction or bleeding disorders;
* Allergic to iodine contrast agent or adenosine, or ineligible for adenosine;
* Participated in other clinical trials within 1 months;
* Other situations that were not suitable for inclusion, as judged by investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stable angina, unstable angina or myocardial infarction after the acute phase
Sampling Method: Probability Sample
Enrollment: 318 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of AccuFFRangio to determine hemodynamically significant coronary artery stenosis compared to FFR as the reference standard | 7 days
  Hemodynamically significant coronary artery stenosis: FFR≤0.8

SECONDARY OUTCOMES:
Sensitivity and specificity of AccuFFRangio to determine hemodynamically significant coronary artery stenosis compared to FFR as the reference standard | 7 days
  Hemodynamically significant coronary artery stenosis: FFR≤0.8
AUC of AccuFFRangio for discrimination of hemodynamically significant coronary artery stenosis | 7 days
  Hemodynamically significant coronary artery stenosis: FFR≤0.8

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang, China

REFERENCES:
- [Derived] Jiang J, Hu Y, Li C, Dong L, Xu J, Tang L, Jiang W, Du C, Jiang X, Lyu Y, Leng X, Li C, Koo BK, Xiang J, Ge J, Wang J. Diagnostic Accuracy of Computational Fluid Dynamics-Based Fractional Flow Reserve Derived From Coronary Angiography: The ACCURATE Study. J Am Heart Assoc. 2025 Jan 7;14(1):e035672. doi: 10.1161/JAHA.124.035672. Epub 2024 Dec 24. PMID 39719423